CLINICAL TRIAL: NCT03991611
Title: Tailored Multicomponent Program for Discomfort Reduction in Critically il Patients May Decrease Post-traumatic Stress Disorder in General ICU Survivors at One Year
Brief Title: Reducing Post-traumatic Stress Disorder After ICU Discharge With the IPREA3 Program
Acronym: PTSD-REA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier of Chartres (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2019-A00151-56
Record Dates: First submitted 2019-06-11; First posted 2019-06-19 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2021-07

CONDITIONS: Critical Illness
Keywords: Critical care; Post-traumatic stress disorder; Discomfort; Tailored program; Patient-reported outcome; ICU; COVID-19
MeSH Terms: conditions — Critical Illness; Stress Disorders, Post-Traumatic; COVID-19

STUDY DESIGN:
Intervention Model Description: Stepped wedge cluster randomized trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- IPREA3 program (Experimental): Application of the IPREA 3 program (multicomponent intervention to reduce perceived discomforts in critically ill patients) for at least 5 months
  Interventions: Other: Administration of the IPREA3 questionnaire; Other: Immediate feedback through electronic reminder messages; Other: Targeted interventions in each ICU to reduce discomforts; Other: 1 year follow-up to assess psychiatric morbidity
- Intermediate group (Other): Application of the IPREA 3 program (multicomponent intervention to reduce perceived discomforts in critically ill patients) for less than 5 months
  Interventions: Other: Administration of the IPREA3 questionnaire; Other: Immediate feedback through electronic reminder messages; Other: Targeted interventions in each ICU to reduce discomforts
- Standard care (Active Comparator): Standard care
  Interventions: Other: Administration of the IPREA3 questionnaire; Other: 1 year follow-up to assess psychiatric morbidity
- PTSD-REA_COVID cohort (Other): ICU admission between March 1, 2020 and April 30, 2020.
  Interventions: Other: 6 months follow-up to assess the prevalence of PTSD symptoms; Other: 1 year follow-up to assess psychiatric morbidity

INTERVENTIONS:
Other: Administration of the IPREA3 questionnaire — On the day of the ICU discharge, the bedside nurse administers to the patient the 18-item IPREA questionnaire i.e the nurse asks the patient to rate from 0 to 10 the severity of each discomfort source contained in the IPREA3 questionnaire experienced during the entire stay in the ICU
  Arms: IPREA3 program; Intermediate group; Standard care
Other: Immediate feedback through electronic reminder messages — After the nurse had administered the questionnaire, warning messages are displayed on the screen corresponding to the key points to prevent the three discomforts reported with the highest scores
  Arms: IPREA3 program; Intermediate group
Other: Targeted interventions in each ICU to reduce discomforts — These targeted interventions are implemented through the coordination of two local champions.
  The central coordination IPREA3 team sends each month to the local champions monthly and cumulative discomfort scores of their unit (overall score of discomfort and scores for each item) and their ranking relative to other units assigned to the interventional arm i.e applying the IPREA3 program.
  The local champions organize monthly meetings with the unit staff to present the results in terms of perceived discomforts measured by the IPREA questionnaire, identify main discomfort sources and actions to be conducted to reduce the discomforts reported with the highest scores in the unit and those that are most easily preventable, and assess the efficacy of already applied measures.
  Arms: IPREA3 program; Intermediate group
Other: 6 months follow-up to assess the prevalence of PTSD symptoms — Psychologist will collect the PCL-5, HAD-S, WHOQOL-BREF, LEC-5 items during the telephone follow-up, 6 months after ICU discharge .
  Arms: PTSD-REA_COVID cohort
Other: 1 year follow-up to assess psychiatric morbidity — Psychologist will collect the PCL-5, HAD-S, WHOQOL-BREF, LEC-5 and CTQ items during the telephone follow-up, 1 year after ICU discharge .
  Arms: IPREA3 program; PTSD-REA_COVID cohort; Standard care

SUMMARY:
Reducing discomfort in the intensive care unit (ICU) should be beneficial to longterm outcomes. This study assesses whether a tailored multicomponent program for discomfort reduction may be effective in reducing post-traumatic stress disorder (PTSD) symptoms at 1-year in general ICU survivors.

The psychiatric morbidity may be increased by the COVID-19 epidemic and its consequences on the healthcare system (patient care, reorganization of French ICUs). The main objective of PTSD-REA_COVID cohort is to assess this psychiatric morbidity 6 months after an ICU stay during the epidemic period.

DETAILED DESCRIPTION:
After carrying out the cluster-randomized controlled IPREA3 study demonstrating that a tailored multicomponent program based on assessment of self-perceived discomfort, feedback to the healthcare teams, and tailored site-targeted measures was effective to decrease self-perceived overall discomfort, we performed the 1-year follow-up of ICUs survivors included in the IPREA3 study to assess psychiatric morbidity at 1 year. Our tailored multicomponent program was also associated with less PTSD at 1 year after ICU discharge. Based on this positive long-term result, this study confirms the need to implement a new strategy for reducing discomfort in the ICU based on such programs.

PTSD-REA is a stepped wedge cluster randomized trial involving 18 ICUs. The exposure will be the implementation of a tailored multicomponent program consisting of assessment of ICU-related self-perceived discomforts, immediate and monthly feedback to the healthcare team, and site-specific tailored interventions. The eligible patients will be exposed vs. unexposed general adult ICU survivors. The prevalence of substantial posttraumatic stress disorder (PTSD) symptoms at 1 year will be assessed by using diagnostic criteria adapted to the new definition of PTSD according to DSM-5.

The current context of the COVID-19 pandemic has considerably disrupted the ICUs organizations as well as the patients care which may lead to increased psychiatric morbidity. In this context, it seems necessary to assess this phenomenon in order to anticipate the consequences on patients but also on the healthcare system. The objectives of the PTSD-REA_COVID cohort are to assess the prevalence of PTSD symptoms, 6 months after ICU stay during COVID-19 epidemic and to compare the psychiatric morbidity at 1 year after an ICU stay during epidemic period and non epidmic period.

ELIGIBILITY:
Inclusion Criteria:

* Patients who survived an ICU stay of at least 3 calendar days
* Affiliation to a social security scheme
* First stay in ICU during current short-term hospitalization
* Patient's oral consent to participate in the PTSD-REA_COVID cohort

Exclusion Criteria:

* Deceased during the ICU stay
* Minors
* Under trusteeship
* Without affiliation to a social security scheme
* Transferred to another ICU
* Already hospitalized in ICU during the current short stay
* Already included in the study
* Limitation and cessation of active treatment
* Advance healthcare directive indicating the refusal of ICU stay
* Irreversible state like diminished cognitive capacity based on the investigator's opinion or not understanding French sufficiently to be questioned (language barrier)
* Subject not consenting to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3312 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Presence of posttraumatic stress disorder (PTSD) symptoms at one year after ICU discharge and 6 months ( PTSD-REA_COVID cohort) | One year after ICU discharge
  PTSD symptoms at one year will be assessed from the PCL-5 which is a 20-item self-report measure that assesses the 20 DSM-5 (Diagnostic and Statistical Manual of Mental Disorders) symptoms of PTSD.
  Each item is rated from 0 "Not at all" to 4 "Extremely". A total symptom severity score (range - 0-80) can be obtained by summing the scores for each of the 20 items.
  A provisional PTSD diagnosis can be made by treating each item rated as 2 = "Moderately" or higher as a symptom endorsed, then following the DSM-5 diagnostic rule which requires at least: 1 B item (questions 1-5), 1 C item (questions 6-7), 2 D items (questions 8-14), 2 E items (questions 15-20).

SECONDARY OUTCOMES:
ICU stay's duration | The day of ICU discharge
Number of days with mechanical ventilation | The day of ICU discharge
Overall score of discomfort assessed from the IPREA3 questionnaire | The day of ICU discharge
The duration of hospital stay after ICU discharge | 6 months ( PTSD-REA_COVID cohort) or 1 year after ICU discharge and
Intrusion Symptom Category B assessed from the PCL-5 (Posttraumatic Stress Disorder Checklist ) (Items 1-5) | 6 months ( PTSD-REA_COVID cohort) and1 year after ICU discharge
  Recurrent or involuntary distressing dreams, memories, thoughts, or feelings related to the traumatic event(s)
Persistent Avoidance Category C assessed from the PCL-5 (Items 6-7) | 6 months ( PTSD-REA_COVID cohort) and1 year after ICU discharge
  Avoidance or efforts to avoid internal or external reminders of the traumatic event(s)
Negative Alterations in Cognitions and Mood Category D assessed from PCL 5 (Items 8-14) | 6 months ( PTSD-REA_COVID cohort) and1 year after ICU discharge
  Persistent and exaggerated negative beliefs about oneself, the world, others, negative mood states, inability to experience positive emotions
Alterations in arousal and reactivity Category E assessed from the PCL-5 (Items 15-20) | 6 months ( PTSD-REA_COVID cohort) and1 year after ICU discharge
  Marked increase in arousal or reactivity such as irritability, hypervigilance, exaggerated startle response, sleep or concentration problems exaggerated startle response
Score of the sub-scale A of the questionnaire HAD-S (Hospital and Anxiety Depression Scale) | 6 months ( PTSD-REA_COVID cohort) and1 year after ICU discharge
  Allowing to estimate the presence of anxious symptoms. The scale HAD contains 14 items rated from 0 to 3. The score of Anxiety ( total A) is obtained by summing items 1-3-5-7-9-11-13 and the depressive dimension (total D) is obtained by summing items 2-4-6-8-10-12-14. The maximal note for each of them is 21.
  8 points is a minimum threshold for determining whether the anxiety is clinically meaningful
Score of the sub-scale D of the questionnaire HAD-S ( Hospital and Anxiety Depression Scale) | 6 months ( PTSD-REA_COVID cohort) and1 year after ICU discharge
  Allowing to estimate the presence of anxious symptoms. The scale HAD contains 14 items rated from 0 to 3. The score of Anxiety ( total A) is obtained by summing items 1-3-5-7-9-11-13 and the depressive dimension (total D) is obtained by summing items 2-4-6-8-10-12-14. The maximal note for each of them is 21.
  8 points is a minimum threshold for determining whether Depression is clinically meaningful
Score obtained from The World Health Organization Quality of Life (WHOQOL-BREF) | 6 months ( PTSD-REA_COVID cohort) and1 year after ICU discharge
  The WHOQOL-BREF measure the following broad domains: physical health, psychological health, social relationships, and environment.
  Each item is rated from 0 to 5. The score of each domain is obtained by summing items then standardized on a scale of 0 (worst quality of life related to health in the dimension explored) to 100 (better quality of liferelated to health in the dimension explored).
Number of emergency stays | 6 months ( PTSD-REA_COVID cohort) and1 year after ICU discharge
  Since ICU discharge
Number of hospitalization | 6 months ( PTSD-REA_COVID cohort) and1 year after ICU discharge
  Since ICU discharge
Number of psychiatric or psychological consultation | 6 months ( PTSD-REA_COVID cohort) and1 year after ICU discharge
  Since ICU discharge
The place of leaving after ICU stay | 6 months ( PTSD-REA_COVID cohort) and1 year after ICU discharge
  Evaluated in population of patients living at home before the ICU stay.
Presence of professional activity | 6 months ( PTSD-REA_COVID cohort) and1 year after ICU discharge
  Evaluated in population of patients with a professional activity before ICU stay

CONTACTS AND LOCATIONS:
Overall Officials: Pierre KALFON, MD PhD, Principal Investigator — CH Chartres
Locations (32):
- France (32):
  - CHU Angers, Angers
  - CHU d'Angers, Angers
  - CH d'Auxerre, Auxerre
  - CH de Blois, Blois
  - Clinique Convert, Bourg-en-Bresse
  - CH Bourges, Bourges
  - Hôpital Louis Pasteur, Chartres
  - CHU de Dijon, Dijon
  - CH de Douai, Douai
  - CH Emile Roux, Le Puy-en-Velay
  - CH de Lens, Lens
  - Hôpital Edouard Herriot, Lyon
  - Hôpital Européen de Marseille, Marseille
  - Hôpital Nord_APHM, Marseille
  - CH de Mâcon, Mâcon
  - CH de l'Agglomération Montargoise, Montargis
  - GHR Mulhouse Sud-Alsace, Mulhouse
  - Clinique Ambroise Paré, Neuilly-sur-Seine
  - Hôpital Pasteur 2_CHU de Nice, Nice
  - Hôpital Saint-Louis_APHP, Paris
  - Gaston Cordier_GH La Pitié-Salpêtrière-Charles Foix_APHP, Paris
  - GH La Pitié-Salpêtrière-Charles Foix_APHP, Paris
  - Husson Mourier_GH La Pitié-Salpêtrière-Charles Foix_APHP, Paris
  - CHU de Poitiers, Poitiers
  - Hôpital privé Claude Galien, Quincy-sous-Sénart
  - CH Victor Provo, Roubaix
  - NCT+ - St Gatien, Saint-Cyr-sur-Loire
  - Nouvel Hôpital Civil_CHU de Strasbourg, Strasbourg
  - Hôpital de Hautepierre_CHU de Strasbourg, Strasbourg
  - Hôpital Sainte Musse, Toulon
  - CHRU de Tours, Tours
  - CH de Troyes, Troyes

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Jones C. Surviving the intensive care: residual physical, cognitive, and emotional dysfunction. Thorac Surg Clin. 2012 Nov;22(4):509-16. doi: 10.1016/j.thorsurg.2012.07.003. Epub 2012 Aug 25. PMID 23084614
- [Result] Jones C, Skirrow P, Griffiths RD, Humphris GH, Ingleby S, Eddleston J, Waldmann C, Gager M. Rehabilitation after critical illness: a randomized, controlled trial. Crit Care Med. 2003 Oct;31(10):2456-61. doi: 10.1097/01.CCM.0000089938.56725.33. PMID 14530751
- [Result] Pacella ML, Hruska B, Delahanty DL. The physical health consequences of PTSD and PTSD symptoms: a meta-analytic review. J Anxiety Disord. 2013 Jan;27(1):33-46. doi: 10.1016/j.janxdis.2012.08.004. Epub 2012 Sep 13. PMID 23247200
- [Result] Pandharipande PP, Girard TD, Jackson JC, Morandi A, Thompson JL, Pun BT, Brummel NE, Hughes CG, Vasilevskis EE, Shintani AK, Moons KG, Geevarghese SK, Canonico A, Hopkins RO, Bernard GR, Dittus RS, Ely EW; BRAIN-ICU Study Investigators. Long-term cognitive impairment after critical illness. N Engl J Med. 2013 Oct 3;369(14):1306-16. doi: 10.1056/NEJMoa1301372. PMID 24088092
- [Result] Davydow DS, Hough CL, Zatzick D, Katon WJ. Psychiatric symptoms and acute care service utilization over the course of the year following medical-surgical ICU admission: a longitudinal investigation*. Crit Care Med. 2014 Dec;42(12):2473-81. doi: 10.1097/CCM.0000000000000527. PMID 25083985
- [Result] Dowdy DW, Eid MP, Dennison CR, Mendez-Tellez PA, Herridge MS, Guallar E, Pronovost PJ, Needham DM. Quality of life after acute respiratory distress syndrome: a meta-analysis. Intensive Care Med. 2006 Aug;32(8):1115-24. doi: 10.1007/s00134-006-0217-3. Epub 2006 Jun 17. PMID 16783553
- [Result] Granja C, Lopes A, Moreira S, Dias C, Costa-Pereira A, Carneiro A; JMIP Study Group. Patients' recollections of experiences in the intensive care unit may affect their quality of life. Crit Care. 2005 Apr;9(2):R96-109. doi: 10.1186/cc3026. Epub 2005 Jan 31. PMID 15774056
- [Result] McKinley S, Aitken LM, Alison JA, King M, Leslie G, Burmeister E, Elliott D. Sleep and other factors associated with mental health and psychological distress after intensive care for critical illness. Intensive Care Med. 2012 Apr;38(4):627-33. doi: 10.1007/s00134-012-2477-4. Epub 2012 Feb 9. PMID 22318635
- [Result] Schelling G, Richter M, Roozendaal B, Rothenhausler HB, Krauseneck T, Stoll C, Nollert G, Schmidt M, Kapfhammer HP. Exposure to high stress in the intensive care unit may have negative effects on health-related quality-of-life outcomes after cardiac surgery. Crit Care Med. 2003 Jul;31(7):1971-80. doi: 10.1097/01.CCM.0000069512.10544.40. PMID 12847391
- [Result] Bienvenu OJ, Gellar J, Althouse BM, Colantuoni E, Sricharoenchai T, Mendez-Tellez PA, Shanholtz C, Dennison CR, Pronovost PJ, Needham DM. Post-traumatic stress disorder symptoms after acute lung injury: a 2-year prospective longitudinal study. Psychol Med. 2013 Dec;43(12):2657-71. doi: 10.1017/S0033291713000214. Epub 2013 Feb 26. PMID 23438256
- [Result] Davydow DS, Gifford JM, Desai SV, Needham DM, Bienvenu OJ. Posttraumatic stress disorder in general intensive care unit survivors: a systematic review. Gen Hosp Psychiatry. 2008 Sep-Oct;30(5):421-34. doi: 10.1016/j.genhosppsych.2008.05.006. Epub 2008 Jul 30. PMID 18774425
- [Result] Jones C, Griffiths RD, Humphris G, Skirrow PM. Memory, delusions, and the development of acute posttraumatic stress disorder-related symptoms after intensive care. Crit Care Med. 2001 Mar;29(3):573-80. doi: 10.1097/00003246-200103000-00019. PMID 11373423
- [Result] Schelling G, Stoll C, Haller M, Briegel J, Manert W, Hummel T, Lenhart A, Heyduck M, Polasek J, Meier M, Preuss U, Bullinger M, Schuffel W, Peter K. Health-related quality of life and posttraumatic stress disorder in survivors of the acute respiratory distress syndrome. Crit Care Med. 1998 Apr;26(4):651-9. doi: 10.1097/00003246-199804000-00011. PMID 9559601
- [Result] Jackson JC, Hart RP, Gordon SM, Hopkins RO, Girard TD, Ely EW. Post-traumatic stress disorder and post-traumatic stress symptoms following critical illness in medical intensive care unit patients: assessing the magnitude of the problem. Crit Care. 2007;11(1):R27. doi: 10.1186/cc5707. PMID 17316451
- [Result] Parker AM, Sricharoenchai T, Raparla S, Schneck KW, Bienvenu OJ, Needham DM. Posttraumatic stress disorder in critical illness survivors: a metaanalysis. Crit Care Med. 2015 May;43(5):1121-9. doi: 10.1097/CCM.0000000000000882. PMID 25654178
- [Result] Patel MB, Jackson JC, Morandi A, Girard TD, Hughes CG, Thompson JL, Kiehl AL, Elstad MR, Wasserstein ML, Goodman RB, Beckham JC, Chandrasekhar R, Dittus RS, Ely EW, Pandharipande PP. Incidence and Risk Factors for Intensive Care Unit-related Post-traumatic Stress Disorder in Veterans and Civilians. Am J Respir Crit Care Med. 2016 Jun 15;193(12):1373-81. doi: 10.1164/rccm.201506-1158OC. PMID 26735627
- [Result] Garrouste-Orgeas M, Coquet I, Perier A, Timsit JF, Pochard F, Lancrin F, Philippart F, Vesin A, Bruel C, Blel Y, Angeli S, Cousin N, Carlet J, Misset B. Impact of an intensive care unit diary on psychological distress in patients and relatives*. Crit Care Med. 2012 Jul;40(7):2033-40. doi: 10.1097/CCM.0b013e31824e1b43. PMID 22584757
- [Result] Cuthbertson BH, Rattray J, Campbell MK, Gager M, Roughton S, Smith A, Hull A, Breeman S, Norrie J, Jenkinson D, Hernandez R, Johnston M, Wilson E, Waldmann C; PRaCTICaL study group. The PRaCTICaL study of nurse led, intensive care follow-up programmes for improving long term outcomes from critical illness: a pragmatic randomised controlled trial. BMJ. 2009 Oct 16;339:b3723. doi: 10.1136/bmj.b3723. PMID 19837741
- [Result] Bergbom-Engberg I, Haljamae H. Patient experiences during respirator treatment--reason for intermittent positive-pressure ventilation treatment and patient awareness in the intensive care unit. Crit Care Med. 1989 Jan;17(1):22-5. doi: 10.1097/00003246-198901000-00006. PMID 2642400
- [Result] Nelson JE, Meier DE, Oei EJ, Nierman DM, Senzel RS, Manfredi PL, Davis SM, Morrison RS. Self-reported symptom experience of critically ill cancer patients receiving intensive care. Crit Care Med. 2001 Feb;29(2):277-82. doi: 10.1097/00003246-200102000-00010. PMID 11246306
- [Result] Novaes MA, Knobel E, Bork AM, Pavao OF, Nogueira-Martins LA, Ferraz MB. Stressors in ICU: perception of the patient, relatives and health care team. Intensive Care Med. 1999 Dec;25(12):1421-6. doi: 10.1007/s001340051091. PMID 10660851
- [Result] Rotondi AJ, Chelluri L, Sirio C, Mendelsohn A, Schulz R, Belle S, Im K, Donahoe M, Pinsky MR. Patients' recollections of stressful experiences while receiving prolonged mechanical ventilation in an intensive care unit. Crit Care Med. 2002 Apr;30(4):746-52. doi: 10.1097/00003246-200204000-00004. PMID 11940739
- [Result] Simini B. Patients' perceptions of intensive care. Lancet. 1999 Aug 14;354(9178):571-2. doi: 10.1016/S0140-6736(99)02728-2. PMID 10470711
- [Result] Soehren P. Stressors perceived by cardiac surgical patients in the intensive care unit. Am J Crit Care. 1995 Jan;4(1):71-6. PMID 7894560
- [Result] Kalfon P, Mimoz O, Auquier P, Loundou A, Gauzit R, Lepape A, Laurens J, Garrigues B, Pottecher T, Malledant Y. Development and validation of a questionnaire for quantitative assessment of perceived discomforts in critically ill patients. Intensive Care Med. 2010 Oct;36(10):1751-1758. doi: 10.1007/s00134-010-1902-9. Epub 2010 May 26. PMID 20502874
- [Result] Kalfon P, Baumstarck K, Estagnasie P, Geantot MA, Berric A, Simon G, Floccard B, Signouret T, Boucekine M, Fromentin M, Nyunga M, Sossou A, Venot M, Robert R, Follin A, Audibert J, Renault A, Garrouste-Orgeas M, Collange O, Levrat Q, Villard I, Thevenin D, Pottecher J, Patrigeon RG, Revel N, Vigne C, Azoulay E, Mimoz O, Auquier P; IPREA Study group. A tailored multicomponent program to reduce discomfort in critically ill patients: a cluster-randomized controlled trial. Intensive Care Med. 2017 Dec;43(12):1829-1840. doi: 10.1007/s00134-017-4991-x. Epub 2017 Nov 27. PMID 29181557
- [Result] Kalfon P, Alessandrini M, Boucekine M, Renoult S, Geantot MA, Deparis-Dusautois S, Berric A, Collange O, Floccard B, Mimoz O, Julien A, Robert R, Audibert J, Renault A, Follin A, Thevenin D, Revel N, Venot M, Patrigeon RG, Signouret T, Fromentin M, Sharshar T, Vigne C, Pottecher J, Levrat Q, Sossou A, Garrouste-Orgeas M, Quenot JP, Boulle C, Azoulay E, Baumstarck K, Auquier P; IPREA-AQVAR Study Group. Tailored multicomponent program for discomfort reduction in critically ill patients may decrease post-traumatic stress disorder in general ICU survivors at 1 year. Intensive Care Med. 2019 Feb;45(2):223-235. doi: 10.1007/s00134-018-05511-y. Epub 2019 Jan 30. PMID 30701294
- [Result] Creamer M, Bell R, Failla S. Psychometric properties of the Impact of Event Scale - Revised. Behav Res Ther. 2003 Dec;41(12):1489-96. doi: 10.1016/j.brat.2003.07.010. PMID 14705607
- [Result] Blevins CA, Weathers FW, Davis MT, Witte TK, Domino JL. The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5): Development and Initial Psychometric Evaluation. J Trauma Stress. 2015 Dec;28(6):489-98. doi: 10.1002/jts.22059. Epub 2015 Nov 25. PMID 26606250
- [Result] Birmes P, Brunet A, Benoit M, Defer S, Hatton L, Sztulman H, Schmitt L. Validation of the Peritraumatic Dissociative Experiences Questionnaire self-report version in two samples of French-speaking individuals exposed to trauma. Eur Psychiatry. 2005 Mar;20(2):145-51. doi: 10.1016/j.eurpsy.2004.06.033. PMID 15797699
- [Result] Jehel L, Brunet A, Paterniti S, Guelfi JD. [Validation of the Peritraumatic Distress Inventory's French translation]. Can J Psychiatry. 2005 Jan;50(1):67-71. doi: 10.1177/070674370505000112. French. PMID 15754668
- [Result] Gray MJ, Litz BT, Hsu JL, Lombardo TW. Psychometric properties of the life events checklist. Assessment. 2004 Dec;11(4):330-41. doi: 10.1177/1073191104269954. PMID 15486169
- [Result] Kubany ES, Haynes SN, Leisen MB, Owens JA, Kaplan AS, Watson SB, Burns K. Development and preliminary validation of a brief broad-spectrum measure of trauma exposure: the Traumatic Life Events Questionnaire. Psychol Assess. 2000 Jun;12(2):210-24. doi: 10.1037//1040-3590.12.2.210. PMID 10887767
- [Result] Bernstein DP, Fink L, Handelsman L, Foote J, Lovejoy M, Wenzel K, Sapareto E, Ruggiero J. Initial reliability and validity of a new retrospective measure of child abuse and neglect. Am J Psychiatry. 1994 Aug;151(8):1132-6. doi: 10.1176/ajp.151.8.1132. PMID 8037246
- [Result] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Result] Baumann C, Erpelding ML, Regat S, Collin JF, Briancon S. The WHOQOL-BREF questionnaire: French adult population norms for the physical health, psychological health and social relationship dimensions. Rev Epidemiol Sante Publique. 2010 Feb;58(1):33-9. doi: 10.1016/j.respe.2009.10.009. Epub 2010 Jan 21. PMID 20096515
- [Derived] Kalfon P, El-Hage W, Geantot MA, Favier C, Bodet-Contentin L, Kuteifan K, Olivier PY, Thevenin D, Pottecher J, Crozon-Clauzel J, Mauchien B, Galbois A, de Varax R, Valera S, Estagnasie P, Berric A, Nyunga M, Revel N, Simon G, Kowalski B, Sossou A, Signouret T, Leone M, Delale C, Seemann A, Lasocki S, Quenot JP, Monsel A, Michel O, Page M, Patrigeon RG, Nicola W, Thille AW, Hekimian G, Auquier P, Baumstarck K; PTSD-REA Study group. Impact of COVID-19 on posttraumatic stress disorder in ICU survivors: a prospective observational comparative cohort study. Crit Care. 2024 Mar 14;28(1):77. doi: 10.1186/s13054-024-04826-1. PMID 38486304